CLINICAL TRIAL: NCT02937194
Title: Family-centered Oral Health Promotion for New Parents and Their Infants: a Randomized Controlled Trial
Brief Title: Family-centered Oral Health Promotion for New Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Government (Other Government); Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Professor May C.M. Wong, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GRF HKU 782213M
Record Dates: First submitted 2016-10-05; First posted 2016-10-18 (Estimated); Results first posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-03

CONDITIONS: Dental Caries
Keywords: Early childhood caries (ECC); Oral health promotion; Randomized controlled trial
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personal oral health instruction + pamphlets distribution (Experimental): Personal oral health instruction (OHI) for the expectant mothers and their husbands together with oral health education materials on infant's tooth development and eruption, establishment of proper feeding, dietary and toothbrushing habits will be given before baby delivery. Reinforcement of OHI and demonstrations on how to clean the infant's oral cavities and perform toothbrushing will be delivered after the babies are born.
  Interventions: Behavioral: Personal oral health instruction + pamphlets distribution
- Pamphlets distribution (Active Comparator): Pamphlets for adults' and pregnant women's oral health care will be distributed when recruited and information on the babies' oral health care will be distributed before baby delivery.
  Interventions: Behavioral: Pamphlets distribution

INTERVENTIONS:
Behavioral: Personal oral health instruction + pamphlets distribution — Personal oral health instruction (OHI) and oral health pamphlets distribution
  Arms: Personal oral health instruction + pamphlets distribution
Behavioral: Pamphlets distribution — Oral health pamphlets distribution
  Arms: Pamphlets distribution

SUMMARY:
Early childhood caries (ECC) is a global health problem that causes pain and infection to the children affected. It is a common disease among preschool children in Hong Kong. There is a great need to improve at-home ECC preventive measures through oral health promotional activities as early as possible to parents.

The investigators will propose a 4-year randomized controlled trial of family-centered oral health promotion for new parents which aims to increase the proportion of parents brushing their infants' teeth at 1 year, establishing proper feeding and dietary habits, reducing the transfer of MS from the parents to their infants and then reducing the risk of ECC of the children at 3 years. The investigators also aim to improve the oral hygiene status of the new parents and prevention of oral diseases among themselves.

First-time expectant mothers and their husbands will be recruited. The recruited families will be randomly allocated to the test and control groups. In the test group, personal hygiene instruction (OHI) for the expectant mothers and their husbands together with oral health education materials on infant's tooth development and eruption, establishment of proper feeding, dietary and toothbrushing habits will be given before the delivery of the new born babies. Reinforcement of OHI and demonstrations on how to clean the infant's oral cavities and perform toothbrushing will be delivered after the babies are born. Comprehensive data will be collected from the mothers, fathers and the infants in both the test and control groups at different time points through dental examination, biological testing and questionnaire survey. The CONSORT statement will be strictly followed when conducting the clinical trial, analyzing the data and reporting the results.

It is anticipated that the effectiveness of oral health promotion starting at the pregnancy period and for both expecting mothers and their husbands will be greater in preventing the infants from developing ECC. Furthermore, establishing good oral health care habits will have long term benefits, helping safeguard the oral health of the children as they grow and the family as a whole. This study will also provide much needed evidence for the further development of oral health policies and oral health promotion programmes in Hong Kong; specifically how these can be integrated into family health education so as to achieve a higher effectiveness. This will contribute significantly to the improvement of oral health in the population of Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* First-time pregnancy
* Of Chinese ethnicity
* Ability to speak Cantonese and read traditional Chinese

Exclusion Criteria:

* Pregnant women with any communication difficulties noted
* Informed consent not obtained

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yu KF, Wen W, Liu P, Gao X, Lo ECM, Wong MCM. Effectiveness of Family-Centered Oral Health Promotion on Toddler Oral Health in Hong Kong. J Dent Res. 2022 Mar;101(3):286-294. doi: 10.1177/00220345211036663. Epub 2021 Sep 13. PMID 34515552
- [Derived] Liu P, Wen W, Yu KF, Gao X, Lo ECM, Wong MCM. Effectiveness of a family-centered behavioral and educational counselling approach to improve periodontal health of pregnant women: a randomized controlled trial. BMC Oral Health. 2020 Oct 16;20(1):284. doi: 10.1186/s12903-020-01265-6. PMID 33066773

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The pregnant women and their husbands were recruited from the Obstetrics & Gynaecology Department of three public hospitals and from two Maternal and Child Health Centers in Hong Kong. The potential participants were approached during their prenatal visits with minimal disturbance to the routine care at the recruitment sites. Written informed consent was obtained from both the pregnant woman and the husband. The recruitment period was from June 2014 to June 2016.
Period: 1-year Followup
Arm/Group | Personal Oral Health Instruction + Pamphlets Distribution | Pamphlets Distribution
Started | 294 | 286
Completed | 223 | 218
Not Completed | 71 | 68
Period: 2-years Followup
Arm/Group | Personal Oral Health Instruction + Pamphlets Distribution | Pamphlets Distribution
Started | 294 (The researchers contacted all the participants recruited/enrolled at baseline at each follow-up regardless if they had participated in the previous follow-up or not. So the number started equals 294 for each follow-up.) | 286 (The researchers contacted all the participants recruited/enrolled at baseline at each follow-up regardless if they had participated in the previous follow-up or not. So the number started equals 286 for each follow-up.)
Completed | 216 | 208
Not Completed | 78 | 78
Period: 3-years Followup
Arm/Group | Personal Oral Health Instruction + Pamphlets Distribution | Pamphlets Distribution
Started | 294 (The researchers contacted all the participants recruited/enrolled at baseline at each follow-up regardless if they had participated in the previous follow-up or not. So the number started equals 294 for each follow-up.) | 286 (The researchers contacted all the participants recruited/enrolled at baseline at each follow-up regardless if they had participated in the previous follow-up or not. So the number started equals 286 for each follow-up.)
Completed | 228 | 208
Not Completed | 66 | 78

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Personal Oral Health Instruction + Pamphlets Distribution | Pamphlets Distribution | Total
Number analyzed (Participants) | 294 | 286 | 580
Age, Continuous [Mean (Standard Deviation); unit: years] — Mother's age
  years | 31.7 (3.7) | 31.6 (4.2) | 31.7 (4.0)
Age, Continuous [Mean (Standard Deviation); unit: years] — Father's age
  years | 33.9 (5.1) | 33.4 (5.2) | 33.6 (5.1)
Sex/Gender, Customized [Number; unit: Families]
  Mother | 294 | 286 | 580
  Father | 294 | 286 | 580
Race/Ethnicity, Customized [Number; unit: Families]
  Chinese | 294 | 286 | 580

OUTCOME MEASURES:

1. Primary Outcome: Early Childhood Caries (ECC)
Description: Prevalence of early childhood caries (ECC) among study children at 36 months
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Personal Oral Health Instruction + Pamphlets Distribution | Pamphlets Distribution
Number analyzed (Participants) | 228 | 208
Participants | 8 | 41

2. Primary Outcome: Parental Toothbrushing on Infants
Description: Proportion of parents who brushed their infants' teeth regularly twice daily at 12 months
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Personal Oral Health Instruction + Pamphlets Distribution | Pamphlets Distribution
Number analyzed (Participants) | 223 | 218
Participants | 74 | 76

3. Secondary Outcome: Feeding Habits on Infants
Description: Proportion of infants falling asleep during milk-feeding
Time Frame: 12 months
Population: The numbers of participants analyzed here are those who finished basiline and one-year follow-up examination.
Measure: Count of Participants; unit: Participants
Arm/Group | Personal Oral Health Instruction + Pamphlets Distribution | Pamphlets Distribution
Number analyzed (Participants) | 218 | 223
Participants | 57 | 63

4. Secondary Outcome: Ratio of Mutans Streptococci (MS)
Description: Proportion of MS with respect to the total bacterial count
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Ratio of MS in the total bacterial count
Arm/Group | Personal Oral Health Instruction + Pamphlets Distribution | Pamphlets Distribution
Number analyzed (Participants) | 216 | 208
Ratio of MS in the total bacterial count | 6.1 (15.7) | 11.6 (17.8)

5. Secondary Outcome: Mothers' Gingival Bleeding
Description: Percentage of probing sites with gingival bleeding (BOP%, range 0-100%)
Time Frame: 12 months
Population: The numbers of participants analyzed here are those who finished basiline and one-year follow-up gingival bleeding examination.
Measure: Mean (Standard Deviation); unit: Percentage of sites with bleeding
Arm/Group | Personal Oral Health Instruction + Pamphlets Distribution | Pamphlets Distribution
Number analyzed (Participants) | 188 | 181
Percentage of sites with bleeding | 35 (29) | 46 (26)

ADVERSE EVENTS:
Time Frame: 1 year, 2 years and 3 years followup
Arm/Group | Personal Oral Health Instruction + Pamphlets Distribution | Pamphlets Distribution
All-Cause Mortality (participants affected / at risk) | 0/294 | 0/286
Serious Adverse Events (participants affected / at risk) | 0/294 | 0/286
Other Adverse Events (participants affected / at risk) | 0/294 | 0/286

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/94/NCT02937194/Prot_SAP_000.pdf